CLINICAL TRIAL: NCT02888067
Title: Surgical Conditions During Vocal Cord Surgery Requiring Jet Ventilation in Patients With Moderate vs. Deep Neuromuscular Block
Brief Title: Surgical Conditions During Vocal Cord Surgery Requiring Jet Ventilation With Moderate vs. Deep Neuromuscular Block
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Thomas Schricker (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Thomas Schricker, Professor and Chairman,Department of Anesthesia, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2017-2754
Record Dates: First submitted 2016-08-12; First posted 2016-09-02 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: High-Frequency Jet Ventilation; Vocal Cord Resection
Keywords: Neuromuscular Blockade
MeSH Terms: interventions — Rocuronium; Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate neuromuscular blockade (MNB) (Active Comparator): The goal is to realize a moderate NMB (TOF 1-2 twitches). NMB will be induced with a bolus dose of rocuronium (Non-depolarizing Skeletal Neuromuscular Blocking Agent). If the target TOF values was not reached bolus doses of rocuronium (5 mg) will be given to achieve the target.
  This represents the standard care in our institution for this type of surgery. At the end of surgery, neuromuscular blockade in all patients will be reversed by sugammadex: patients in the moderate neuromuscular blockade group will receive sugammadex (Selective Relaxant Binding Agent).
  Interventions: Drug: Rocuronium bromide 0.5 mg/kg; Drug: Sugammadex sodium 2 mg/kg
- Deep neuromuscular blockade (MNB) (Active Comparator): The goal is to realize a deep MNB (TOF zero twitches). NMB will be induced with a bolus dose of rocuronium (Non-depolarizing Skeletal Neuromuscular Blocking Agent). If the target TOF values was not reached bolus doses of rocuronium (5 mg) will be given to achieve the target.
  At the end of surgery, neuromuscular blockade in all patients will be reversed by sugammadex: patients in the deep neuromuscular blockade group will receive sugammadex (Selective Relaxant Binding Agent).
  Interventions: Drug: Rocuronium bromide 1.0 mg/kg; Drug: Sugammadex sodium 4 mg/kg

INTERVENTIONS:
Drug: Rocuronium bromide 0.5 mg/kg — Moderate neuromuscular blockade with rocuronium bromide
  Other Names: Zemuron®
  Arms: Moderate neuromuscular blockade (MNB)
Drug: Rocuronium bromide 1.0 mg/kg — Deep neuromuscular blockade with rocuronium bromide
  Other Names: Zemuron®
  Arms: Deep neuromuscular blockade (MNB)
Drug: Sugammadex sodium 2 mg/kg — Reversal with sugammadex sodium
  Other Names: Bridion™
  Arms: Moderate neuromuscular blockade (MNB)
Drug: Sugammadex sodium 4 mg/kg — Reversal with sugammadex sodium
  Other Names: Bridion™
  Arms: Deep neuromuscular blockade (MNB)

SUMMARY:
The purpose of this study is to determine whether deep neuromuscular blockade provides better surgical conditions than moderate neuromuscular blockade in patients undergoing vocal cord resections requiring jet ventilation.

DETAILED DESCRIPTION:
To optimize anatomical exposure and to minimize direct manipulation of local lesions endotracheal intubation often is avoided in patients undergoing vocal cord surgery.

Instead intermittent so called jet ventilation is carried out by using the Hunsaker Mon-jet tube. The safe conduct of these procedures requires full muscle paralysis. In clinical practice, however, deep neuromuscular blockade (NMB) usually cannot be established for this relatively short surgery (<1h) because of an increased risk of prolonged NMB and postoperative ventilation.

The novel neuromuscular blockade reversal agent sugammadex may prove particularly useful in this patient population because it allows fast and reliable reversal of even deep NMB. Deeper muscle paralysis during vocal cord surgery may be associated with better surgical conditions.

The purpose of this study is to determine whether deep neuromuscular blockade provides better surgical conditions than moderate neuromuscular blockade in patients undergoing vocal cord resections requiring jet ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Elective vocal cord resection with an expected length of the procedure longer than 20 minutes and requiring jet ventilation

Exclusion Criteria:

* Patients younger than 18 years old
* Patients unable to give written informed consent
* Patients with known or suspected neuromuscular disease
* Patients with allergies to medications to be used during anesthesia
* Patients with a (family) history of malignant hyperthermia
* Patients with renal insufficiency (serum creatinine >2 times normal or a glomerular filtration rate <60 ml/h)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Five-point surgical rating scale (SRS) | during surgery, an average period of 50 minutes
  Surgical conditions during surgery will be assessed by the surgeon using a five-point surgical rating scale at 10 minutes intervals

SECONDARY OUTCOMES:
Drug dosages | Through study completion, an average of 4 hours
  Drugs and dosages used during the study
Time to extubation | During the stay in the operation room, an average of 60 minutes
  Time from reversal to optimal extubation conditions (TOF ratio <0.9)
Heart rate | During the stay in the operation and recovery room, an average of 4 hours
Arterial blood pressure | During the stay in the operation and recovery room, an average of 4 hours
Oxygen saturation | During the stay in the operation and recovery room, an average of 4 hours
Respiratory rate | During the stay in the operation and recovery room, an average of 4 hours
Body temperature | During the stay in the operation and recovery room, an average of 4 hours
Duration of surgery | During the stay in the operation room, an average of 50 minutes
Duration of post-anesthesia care unit (PACU) stay | During the stay in the recovery room, an average of 3 hours
  Time spent in the PACU
Pain score | During the stay in the operation and recovery room, an average of 4 hours
  On an 11-point numerical rating scale from 0 = no pain, to 10 = most severe pain imaginable at PACU
Occurence of nausea/vomiting | During the stay in the operation and recovery room, an average of 4 hours
Sedation | During the stay in the operation and recovery room, an average of 4 hours
  On a five-point scale ranging from 0 = normal alertness to 5 = not aroused by a painful stimulus at PACU

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schricker, M.D., PhD., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- MUHC, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No